CLINICAL TRIAL: NCT04945395
Title: The Effect of Using Functional Electric Stimulation for the Recovery of Dorsiflexion During Rehabilitation of Gait Function, in the Subacute Phase After Stroke- a Randomized Controlled Exploratory Study
Brief Title: Effect of Functional Electric Stimulation for Recovery of Dorsiflexion After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: KTH Royal Institute of Technology (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, PhD, Reg Physiotherapist, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FES-study
Record Dates: First submitted 2021-06-03; First posted 2021-06-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Stroke; Ambulation Difficulty; Hemiplegia
Keywords: Rehabilitation; Functional electrical stimulation; Walking; Stroke
MeSH Terms: conditions — Stroke; Mobility Limitation; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to the patients´ allocation in terms of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES and conventional training (Experimental): The experimental group will wear the Functional electrical stimulation system L3100 Go for dorsiflexion of the ankle during conventional rehabilitation interventions involving the lower extremity led or instructed by a physiotherapist.
  Interventions: Device: FES and Conventional training
- AFO and Conventional training only (Active Comparator): The control group will wear an ankle-foot-orthosis (AFO) to enhance dorsiflexion of the foot while taking part in conventional rehabilitation interventions involving the lower extremity led or instructed by a physiotherapist.
  Interventions: Device: AFO and Conventional training

INTERVENTIONS:
Device: FES and Conventional training — The experimental group will be fitted with the Functional electrical stimulation system L300 Go to be used during 4 weeks of inpatient rehabilitation in the subacute phase after hemiplegic stroke. Settings will be adjusted continuously to enhance dorsiflexion of the affected foot during walking and mobility training.
  Arms: FES and conventional training
Device: AFO and Conventional training — The control group will be fitted with an ankle-foot-orthosis (AFO) according to clinical practice to enhance dorsiflexion of the foot while taking part in conventional rehabilitation interventions during 4 weeks of inpatient rehabilitation including walking and mobility training in the subacute phase after hemiplegic stroke
  Arms: AFO and Conventional training only

SUMMARY:
The purpose of this project is to investigate the effect of functional electrical stimulation (FES) for recovery of dorsiflexion after stroke. It will be led from the University Department of Rehabilitation Medicine at Danderyd Hospital (RMDS) in collaboration with the MoveAbility Lab at KTH Royal Institute of Technology. Patients referred to RMDS for inpatient rehabilitation early after hemiparetic stroke will be included.

The overall aim is to explore how 4 weeks of training incorporating the FES-system (L300 Go System ® Bioness, Ottobock) effect function of the lower extremity, gait function and mobility when compared to conventional training only, in the subacute stage after stroke.

DETAILED DESCRIPTION:
Participants will be included and allocated to either experimental group with training incorporating the FES-system and conventional training or to control group with conventional training only. Data will be collected before and after the intervention at RMDS and at the MoveAbility Lab. Physical tests and self-scored questionnaires of self-perceived aspects of functioning and disability will be performed at RMDS and gait analysis with 3D cameras and assessment of muscle function with EMG will be performed at the MoveAbilityLab. In addition, a short assessment of body function and activity will be performed weekly at RMDS by the therapist responsible for the rehabilitation intervention.

The experimental group will wear the FES-system L300 Go at all times when the patient is taking part in rehabilitation interventions involving the lower extremity led or instructed by a physiotherapist. The settings will be adjusted by the employee from the technical company and/or the physiotherapist continuously during the intervention if needed. The system will register the distance and time accomplished during each session. Due to risk of skin irritation, if the system is overused in the beginning the experimental group will have access to an ankle-foot-orthosis too.

The control group will wear an ankle-foot-orthosis (AFO) and receive conventional training. The control group will wear a FES-system too, to record the distance and time accomplished during each session, but the system will not be active for stimulation.

ELIGIBILITY:
Eligible will be patients who have suffered a stroke, verified by CT or MRI examination and are admitted to inpatient care at the University Department of Rehabilitation Medicine Stockholm, Danderyd Hospital in Sweden where approximately 220 patients are treated annually (Stroke (50%)).

Inclusion criteria:

* 20 participants with hemiplegia
* Dependence in ambulation (0- 4 according to the Functional Ambulation Categories)
* >= 50 points on the Trunc Control Test.
* Impaired dorsiflexion manifested as impaired voluntarily dorsiflex and to hold the ankle in a dorsiflexed position while sitting and for ambulatory participants: during swing phase and heel strike while walking as demonstrated by visual inspection during gait analysis performed by the physiotherapist.
* Recommended to be fitted with an ankle-foot orthosis (AFO) by an experienced physiotherapist.
* Able to understand study information and to give informed consent.

Exclusion Criteria:

* Contracture severely restricting gait movements at any lower limb joint
* Cardiovascular or other somatic condition incompatible with intensive gait training
* Notifiable infectious disease, contagious infections (e.g. Methicillin Resistant Staphylococcus Aureus (MRSA) or Extended Spectrum Beta Lactamase bacteria (ESBL)). - Not able to participate in the rehabilitation intervention due to behavioral disorder or psychiatric disease.
* The FES-system L300 Go ® should not be used if a the patient has a pacemaker, defibrillator or any electrical implant, a metallic implant in the affected leg, a cancerous lesion in the affected leg, a fracture or dislocation in the affected leg or if the affected leg is swollen, infected, or has inflamed areas or skin eruptions, such as phlebitis, thrombophlebitis, and varicose veins in the affected leg or if the patient is pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Gait Profile Score (GPS) | At baseline and after completion of the 4 week intervention to assess change.
  GPS is a single index measure that summarises the overall deviation of kinematic gait data relative to normative data. The GPS can be decomposed to provide the Gait Variable Score (GVS) (an index that measures single gait variable deviation), for nine key relevant kinematic variables. A larger GPS indicates greater deviation from normal gait
Ankle Sagittal range (degrees) | At baseline and after completion of the 4 week intervention to assess change.
  Assesses range of motion in the ankle (plantarflexion from 0-50 degrees, dorsiflexion from 0-20 degrees)
Ankle Positive work | At baseline and after completion of the 4 week intervention to assess change.
  Assesses the force at the ankle joint (J/kg) detected in gait laboratory
Step length | At baseline and after completion of the 4 week intervention to assess change.
  Step length will be assessed in the gait laboratory with 3D gait analyses
6 minutes walk test | At baseline and after completion of the 4 week intervention to assess change.
  Assesses walking endurance in meters walked
Rated Perceived Exertion (RPE) Scale | At baseline and after completion of the 4 week intervention to assess change.
  Ratings (min 6, max 20) according to the RPE scale are made at the end of the 6 minutes walk test. A higher score indicates a higher degree of perceived exertion.

SECONDARY OUTCOMES:
The Montreal Cognitive Assessment (MoCa) | At baseline and after completion of the 4 week intervention to assess change.
  Assesses mental function (0p max impairment summed up to 30p no detected impairment)
Fugl-Meyer score (FMA-LE) | At baseline, weekly during the intervention and after completion of the 4 week intervention to assess change.
  Assesses sensory and movement related functions in the lower extremity (0p max impairment summed up to 86p max no detected impairment)
Neuroflexor | At baseline, weekly during the intervention, and after completion of the 4 week intervention to assess change.
  Medical technology device. Assesses spasticity by identifying the neural, viscous and elastic components during passive movement using a biomechanical algorithm (presented in Newton)
Modified Ashworth scale 0-5 | At baseline, weekly during the intervention and after completion of the 4 week intervention, to assess change.
  Assesses spasticity on a 6 point scale/muscle (0p no impairment, 5p max impairment/muscle)
Passive range of motion in the lower extremity | At baseline, weekly during the intervention and after completion of the 4 week intervention to assess change.
  Clinical assessment of range of motion with a goniometer
Medical Research Council scale | At baseline and after completion of the 4 week intervention
  Assesses muscle strength on a 6 point scale/muscle (0p max impairment summed up to 5p no impairment/muscle)
The Balance evaluation systems test (BEST-test) | At baseline, weekly during the intervention and after completion of the 4 week intervention to assess change.
  Assesses postural control, incorporating bio-mechanical systems, limits of stability, anticipatory postural adjustment, automatic postural responses, sensory orientation, stability in gait (0p max impairment summed up to 108p no impairment)
The 10 meter walk test | At baseline, weekly during the intervention and after completion of the 4 week intervention to assess change.
  Assesses gait speed
6 minutes walk test | At baseline, weekly during the intervention and after the intervention to assess change
  Assesses walking endurance in meters walked
Rated Perceived Exertion (RPE) Scale | At baseline, weekly during the intervention and after the intervention to assess change
  Ratings (min 6, max 20) according to the RPE scale are made at the end of the 6 minutes walk test.
Indirect Calorimetries | At baseline and after the intervention to assess change
  To assess energy expenditure based on respiratory gas exchange. Will be performed during the 6 minutes walk test.
Electromyography (EMG) | At baseline and after completion of the 4 week intervention to assess change.
  EMG is used to measure muscle activation patterns during gait.
Walking impact scale (MSWS-12 S) | At baseline and after completion of the 4 week intervention to assess change.
  Assesses self-perceived limitations in walking (12p no impairments summed up to 60p max impairment)
The Functional Ambulation Categories (FAC) | At baseline, weekly during the intervention and after completion of the 4 week intervention to assess change.
  Assesses independence in walking (0p nonfunctional, 5p independent) Total score 0-5p
Falls Efficacy Scale (FES-S) | At baseline and after completion of the 4 week intervention to assess change.
  Assesses self perceived balance in every day life activities rated on a 11 point scale (0p not safe at all 10p completely safe). Total score: 0- 130 p
Barthel Index | At baseline, weekly during the intervention and after completion of the 4 week intervention to assess change.
  Assesses independence in mobility and personal care (0p dependent 10/15p independent) Total score 0-100p
Eq-5d-5l | At baseline and after completion of the 4 week intervention to assess change.
  Assesses self perceived health related quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and on a vertical visual analogue scale. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension (1 = no problem, 5 = extreme problems). The vertical visual analogue scale is graded from 0-100 (0 = the worst health you can imagine 100 = the best health you can imagine).
A study specific questionnaire - a questionnaire for the experimental group | After completion of the 4 week intervention
  A questionnaire with 11 questions assessing the patients experience of participating in the study and the use of the FES-system. The patient rates on a 10 graded scale (0 = not at all, 10 = very much): the information given about the study, the experience, usability and comfort of using the system, eventual pain, skin problems and technical problems with the system and experience of eventual benefits from having used the system.
Distance accomplished during each training session | Daily during the intervention
  The FES-system will collect this data to assess training intensity
Time accomplished during each training session | Daily during the intervention
  The FES-system will collect this data to assess training intensity

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Palmcrantz, PhD, Principal Investigator — Dep of Clinical Sciences, Karolinska Institutet
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County, Sweden